

Tel: 01772 522774

Royal Preston Hospital, Sharoe Green Lane, Fulwood, Preston. PR2 9HT

Date:

Centre Number: RPH Study Number: Pilot

Patient Identification Number for this trial:

## **CONSENT FORM Patient version**

Title of Project: Is trans-laryngeal ultrasound (TLUS) a useful tool to evaluate the vocal fold movement abnormalities seen in Inducible Laryngeal Obstruction (ILO) a pilot study.

Name of Researcher: Claire Slinger, Consultant speech & language therapist

| | | | Please initial box |
|---|---|---|---|
| 1. I confirm that I have read and (version 3.0) for the above study ask questions and have had the | . I have had the opportunity to c | | |
| 2. I understand that my participa without giving any reason, witho | | | |
| 3. I understand that relevant sec<br>may be looked at by individuals<br>where it is relevant to my taking<br>individuals to have access to my | dy, | | |
| 4. I agree to take part in the abo | ve study. | | |
| Name of Patient | <br>Date | Signature | |

IRAS Project ID: 298631



| Name of Person | Date | Signature |
|----------------|------|-----------|
| taking consent | | |

When completed: 1 for participant; 1 for researcher site file; 1 (original) to be kept in medical notes.